CLINICAL TRIAL: NCT03692338
Title: INTERVAL: Ipilimumab and Nivolumab Combination Therapy: A Study of a Supervised or Semi-Supervised Exercise InteRVention or Usual Care With Functional Capacity and Quality of Life Evaluations in Subjects With Advanced or Metastatic RenAL Cell Carcinoma
Acronym: INTERVAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Duke University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00082941
Record Dates: First submitted 2018-09-25; First posted 2018-10-02 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: metastatic renal cell carcinoma; ipilimumab; nivolumab; exercise
MeSH Terms: conditions — Carcinoma, Renal Cell; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to one of three cohorts: Supervised exercise, semi-supervised exercise or usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 12 week supervised exercise program (Experimental): Patients will be asked to complete 3 30-minute supervised exercise sessions/week under the guidance of the study exercise physiologist. The preferred mode will be treadmill walking, however, alternatives such as cycling or stair climbing machines will be used. For these sessions, patients will be asked to wear a heart rate monitor. Following a 5 minute warm-up, the exercise physiologist will increase speed to correspond with an intensity of approximately 80% VO2peak for 1-minute before returning to a lower speed for 1-minute (50% VO2peak). Patients will complete up to 20 of each 1-minute interval, then cool-down for 5 minutes. At the end of each higher intensity interval patients will be asked to rate their perceived exertion (RPE).
  Additionally, patients will receive standard of care nivolumab (3 mg/kg i.v.) and ipilimumab (1 mg/kg i.v.) q3 weeks x 4 doses followed by nivolumab at 3 mg/kg q2 weeks.
  Interventions: Behavioral: Exercise
- 12 week semi-supervised exercise program (Experimental): This cohort will complete 12 weeks of a semi-supervised exercise program independently. Patients will be scheduled for an exercise session with a study exercise physiologist during clinical appointments to complete a sample intensity and time specific exercise session. The preferred mode will be walking, however cycling is also permitted. For each session the patient will wear a heart rate monitor. Following a 5 minute warm-up, patients will increase the intensity of exercise to reach a heart rate corresponding to approximately 60% VO2peak, and will continuously maintain this intensity for their individualized duration to elicit the desired energy expenditure. Each week, the exercise physiologist will call the patient and discuss how to approach the next set of exercise sessions.
  Additionally, patients will receive standard of care nivolumab (3 mg/kg i.v.) and ipilimumab (1 mg/kg i.v.) q3 weeks x 4 doses followed by nivolumab at 3 mg/kg q2 weeks.
  Interventions: Behavioral: Exercise
- Control cohort (No Intervention): Participants will have routine care for 12 weeks. This will consist of nivolumab (3 mg/kg i.v.) and ipilimumab (1 mg/kg i.v.) q3 weeks x 4 doses followed by nivolumab at 3 mg/kg q2 weeks.

INTERVENTIONS:
Behavioral: Exercise — Patients will be asked to complete 3 x 30 minute exercise sessions each week.
  Arms: 12 week semi-supervised exercise program; 12 week supervised exercise program

SUMMARY:
This study aims to report the effects of immediate or delayed exercise training on patients with advanced or metastatic renal cell carcinoma who are receiving nivolumab and ipilimumab.

DETAILED DESCRIPTION:
Exercise interventions also have been shown to improve both cancer- and treatment-related fatigue and quality of life across multiple tumor types. Thus, an exercise intervention could improve the tolerability of combination immunotherapy. Furthermore, functional capacity and/or amount of physical activity are associated with survival in several cancers. Finally, there is emerging evidence that exercise training may augment beneficial cancer-specific immune function. This study will examine parallel groups of supervised or semi-supervised exercise training or usual care in patients with mRCC treated with nivolumab and ipilimumab combination therapy. Fitness level will be evaluated by cardiopulmonary exercise testing (CPET), wearable exercise tracking devices and questionnaires after 12 weeks of semi-supervised, home-based exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Scheduled to receive ipilumab and nivolumab as first line of immune checkpoint inhibitor therapy for Renal Cell Carcinoma (RCC).

   a. Patient may receive the first infusion of ipilimumab/nivolumab prior to eligibility determination
3. Subjects with brain metastases are allowed if they are asymptomatic, without edema, and not on greater than or equal to 10mg daily dose of systemic corticosteroids or receiving radiation therapy for at least 14 days prior to beginning protocol therapy.
4. Karnofsky Performance Status (KPS) of at least 70%
5. Able to walk on a treadmill per patient report.
6. Ability to understand English and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Major surgery (e.g. nephrectomy) less than 28 days prior to the first dose of ipilimumab/nivolumab.
2. History of cerebrovascular accident including transient ischemic attack (TIA) within the past 6 months.
3. Osseous metastatic disease with unacceptable risk of impending fracture due to study assessments, in the opinion of the investigator. Note: This criterion must be met prior to CPET.
4. Absolute contraindications to cardiopulmonary exercise testing and/or aerobic training, as determined by the attending oncologist:

   * Uncontrolled arrhythmia causing symptoms or hemodynamic compromise
   * Recurrent syncope
   * Active endocarditis
   * Acute myocarditis or pericarditis
   * Symptomatic severe aortic stenosis
   * Uncontrolled heart failure
   * Acute (within 3 months) pulmonary embolus or pulmonary infarction
   * Thrombosis of lower extremities
   * Suspected dissecting aneurysm
   * Uncontrolled asthma
   * Pulmonary edema
   * Room air desaturation at rest <85%
   * Respiratory failure
   * Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis)
   * Mental impairment leading to inability to cooperate.
   * Poorly controlled hypertension [defined as systolic blood pressure (SBP) of >150 mmHg or diastolic blood pressure (DBP) of >90 mmHg].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Change in Cardiopulmonary function | Baseline, 13 weeks
  Change in VO2 peak

SECONDARY OUTCOMES:
Patient-reported fatigue as measured by the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue scale | 13 weeks
  The FACIT-F measures severity and impact of fatigue on functioning and health-related quality of life experienced in past seven days using 40 statements that patients are asked to rate as 0-4 with 0 being "Not at all" and 4 being "Very much".
Patient-reported activity as measured by the Godin Leisure Time Exercise Questionnaire | 13 weeks
  The Godin Leisure is a patient-reported outcome tool to measure activity
Patient-reported symptoms as measured by the Functional Assessment of Cancer Therapy-Kidney Symptom Index-19 (FKSI-19) | 13 weeks
  The FKSI-19 is a patient-reported outcome tool to measure symptoms of Cancer
Patient health outcome as measured by the EQ-5D health questionnaire | 13 weeks
  The EQ-5d is a patient-reported outcome tool to measure health
Patient-reported activity as measured by the Stanford Brief Activity Survey | 13 weeks
  The Stanford Brief Activity Survey is a patient-reported outcome tool to measure activity
Patient-reported activity as measured by the Incidental and Planned Activity Questionnaire | 13 weeks
  The Incidental and Planned Activity Questionnaire is a patient-reported outcome tool to measure activity

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harrison, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No